CLINICAL TRIAL: NCT04998578
Title: Comparison Of Aesthetic Techniques For Rejuvenation Of Genital Region: A Randomized Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro de Atenção ao Assoalho Pélvico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Caap
Record Dates: First submitted 2019-06-26; First posted 2021-08-10 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Laxity; Skin; Skin Hyperpigmentation; Needlestick Puncture
Keywords: microneedling; laxity; Skin Hyperpigmentation
MeSH Terms: conditions — Cutis Laxa; Hyperpigmentation

STUDY DESIGN:
Intervention Model Description: Group A will only perform microneedling; group B will perform microneedling associated with the use of cosmetic in the office; group C will perform microneedling associated with the cosmetology of office and home use; and group D will perform non-ablative radiofrequency. Due to the application characteristics of the microneedle technique, there is no way to use a placebo group.
Who Masked: Investigator
Masking Description: the data of the participants will be collected by evaluators blind to the study and who will not know the allocation of the patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Microneedling- Group A (Active Comparator): Participants will only perform microneedling
  Interventions: Device: Comparison of aesthetic techniques
- Microneedling and outpatient Cosmetics- Group B (Active Comparator): Microneedling associated with the use of outpatient cosmetics
  Interventions: Device: Comparison of aesthetic techniques
- microneedling and home use cosmetics - Group C (Active Comparator): Microneedling associated with home use cosmetics
  Interventions: Device: Comparison of aesthetic techniques
- Non-ablative radiofrequency - Group D (Active Comparator): Participants will perform only non-ablative radiofrequency
  Interventions: Device: Comparison of aesthetic techniques

INTERVENTIONS:
Device: Comparison of aesthetic techniques — Comparison of aesthetic techniques for rejuvenation and glazing of the genital region

SUMMARY:
The microneedle is a minimally invasive technique, consists of the application of a roller surrounded by small and thin needles that pierce the skin and generate a mechanical stimulus with no ablative effect on the skin. The study aims to test the hypothesis that the technique of microneedle in the treatment of tissue flaccidity and hyperchromia of female external genitalia is safe and with a more effective result in clinical improvement through genital rejuvenation and unification of skin tone when compared to non-ablative radiofrequency technique.

DETAILED DESCRIPTION:
Dissatisfaction with the genital image has been receiving more attention in recent years and is influenced by mediation and the methods of waxing modernity. In the face of this, the number of women in search for aesthetic female genital surgeries. Since the year 2015, the implementation of the Labiaplasty surgery had a growth of 45% worldwide. Brazil is a leader in the procedure, with a total of 23,155 procedures in the year 2016 (ISAPS DATA). However, the Most genital surgical cases are performed unnecessarily, without long-term term, according to a conflict of interest arising from financial gain, generating ethical complications The search for aesthetic non-invasive genital treatments, in its majority, is related to sagging big lips and genital hyperchromia. In the literature, the non-invasive therapeutic resource and with fewer adverse effects described for aesthetics of the genital region is the use of the radiofrequency apparatus ablative, considered to be a safe and effective technique for flaccidity of the cutaneous tissue. It is not described in the literature treatments used for genital hyperchromia, however, several formulations for clearings using Kojic acid and Niacinamide, already described as effective for other regions, are available for marketing primarily for genital year whitening.

Minimally invasive technique, consists of the application of a roller surrounded by small and thin needles that pierce the skin and generate a mechanical stimulus with no ablative effect on the skin.

ELIGIBILITY:
Inclusion Criteria:

• Women aged 18-65 years with skin flaccidity and genital hyperchromia

Exclusion Criteria:

* Patients who use cosmetics in the genital region
* Use of anticoagulant medication
* Use of pacemakers
* Pregnancy
* Dermatoses in the region to be treated and / or local inflammatory condition, without diagnosis of infection
* Difficulty in understanding the proposed instruments

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
External genital Laxity | 1, 3, 6 and 12 months after treatment
  It will be evaluated by turgor, number of skinfolds, evidenced by self report, comparison of images taken before and after the procedure and satisfaction of the patient, verified in the Likert scale and Visual Analog Scale.
Genital Hyperchromia | 1, 3, 6 and 12 months after treatment
  It will be evaluated the uniformity of the skin tone, evidenced by the self report, comparison of images taken before after the procedure and satisfaction of the participant, verified in the scale of Likert and Scale Visual Analog.

SECONDARY OUTCOMES:
Sexual function | 1, 3, 6 and 12 months after treatment
  It will be evaluated through the questionnaire Sexual Quotient - Female Version (QS-F), Female Sexual Function Index (FSFI)
Female Genital Self-Image | 1, 3, 6 and 12 months after treatment
  It will be evaluated through the Female Genital Self-Image Scale (FGSIS) > 26
Melasma Quality of Life | 1, 3, 6 and 12 months after treatment
  It will be evaluated through the Melasma Quality of Life Scale (MELASQoL).

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Centro de Atenção ao Assoalho Pelvico, Salvador, Estado de Bahia
  - Centro de Atenção ao assoalho pélvico, Salvador, Estado de Bahia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vieira-Baptista P, Marchitelli C, Haefner HK, Donders G, Perez-Lopez F. Deconstructing the genitourinary syndrome of menopause. Int Urogynecol J. 2017 May;28(5):675-679. doi: 10.1007/s00192-017-3295-6. Epub 2017 Mar 14. PMID 28293790
- [Background] Marnach ML, Torgerson RR. Vulvovaginal Issues in Mature Women. Mayo Clin Proc. 2017 Mar;92(3):449-454. doi: 10.1016/j.mayocp.2016.10.031. PMID 28259230
- [Background] Filippini M, Del Duca E, Negosanti F, Bonciani D, Negosanti L, Sannino M, Cannarozzo G, Nistico SP. Fractional CO2 Laser: From Skin Rejuvenation to Vulvo-Vaginal Reshaping. Photomed Laser Surg. 2017 Mar;35(3):171-175. doi: 10.1089/pho.2016.4173. Epub 2016 Dec 30. PMID 28056209
- [Background] Portman DJ, Gass ML; Vulvovaginal Atrophy Terminology Consensus Conference Panel. Genitourinary syndrome of menopause: new terminology for vulvovaginal atrophy from the International Society for the Study of Women's Sexual Health and the North American Menopause Society. Menopause. 2014 Oct;21(10):1063-8. doi: 10.1097/GME.0000000000000329. PMID 25160739
- [Background] Lapii GA, Yakovleva AY, Neimark AI. Structural Reorganization of the Vaginal Mucosa in Stress Urinary Incontinence under Conditions of Er:YAG Laser Treatment. Bull Exp Biol Med. 2017 Feb;162(4):510-514. doi: 10.1007/s10517-017-3650-0. Epub 2017 Feb 27. PMID 28243906
- [Background] Ho D, Kraeva E, Wun T, Isseroff RR, Jagdeo J. A single-blind, dose escalation, phase I study of high-fluence light-emitting diode-red light (LED-RL) on human skin: study protocol for a randomized controlled trial. Trials. 2016 Aug 2;17:385. doi: 10.1186/s13063-016-1518-7. PMID 27484782
- [Background] Miyata S, Miyaji H, Kawasaki H, Yamamoto M, Nishida E, Takita H, Akasaka T, Ushijima N, Iwanaga T, Sugaya T. Antimicrobial photodynamic activity and cytocompatibility of Au25(Capt)18 clusters photoexcited by blue LED light irradiation. Int J Nanomedicine. 2017 Apr 4;12:2703-2716. doi: 10.2147/IJN.S131602. eCollection 2017. PMID 28435253
- [Background] Takada A, Matsushita K, Horioka S, Furuichi Y, Sumi Y. Bactericidal effects of 310 nm ultraviolet light-emitting diode irradiation on oral bacteria. BMC Oral Health. 2017 Jun 6;17(1):96. doi: 10.1186/s12903-017-0382-5. PMID 28587675
- [Background] Arunkalaivanan A, Kaur H, Onuma O. Laser therapy as a treatment modality for genitourinary syndrome of menopause: a critical appraisal of evidence. Int Urogynecol J. 2017 May;28(5):681-685. doi: 10.1007/s00192-017-3282-y. Epub 2017 Feb 2. PMID 28154914
- [Background] Nilsson K, Risberg B, Heimer G. The vaginal epithelium in the postmenopause--cytology, histology and pH as methods of assessment. Maturitas. 1995 Jan;21(1):51-6. doi: 10.1016/0378-5122(94)00863-3. PMID 7731384
- [Background] Flores SA, Hall CA. Atrophic Vaginitis(Archived). 2025 Jun 19. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK564341/ PMID 33232011
- [Background] Herbenick D, Reece M. Development and validation of the female genital self-image scale. J Sex Med. 2010 May;7(5):1822-30. doi: 10.1111/j.1743-6109.2010.01728.x. Epub 2010 Mar 3. PMID 20233278
- [Background] Cain JM, Iglesia CB, Dickens B, Montgomery O. Body enhancement through female genital cosmetic surgery creates ethical and rights dilemmas. Int J Gynaecol Obstet. 2013 Aug;122(2):169-72. doi: 10.1016/j.ijgo.2013.03.020. Epub 2013 Jun 2. PMID 23735570
- [Background] McPencow AM, Guess MK. Giving female genital cosmetic surgery a facelift. Maturitas. 2012 Apr;71(4):313-4. doi: 10.1016/j.maturitas.2012.01.012. Epub 2012 Feb 14. No abstract available. PMID 22341089
- [Background] Doddaballapur S. Microneedling with dermaroller. J Cutan Aesthet Surg. 2009 Jul;2(2):110-1. doi: 10.4103/0974-2077.58529. PMID 20808602
- [Background] Ramaut L, Hoeksema H, Pirayesh A, Stillaert F, Monstrey S. Microneedling: Where do we stand now? A systematic review of the literature. J Plast Reconstr Aesthet Surg. 2018 Jan;71(1):1-14. doi: 10.1016/j.bjps.2017.06.006. Epub 2017 Jun 17. PMID 28690124
- [Background] Fabbrocini G, De Vita V, Fardella N, Pastore F, Annunziata MC, Mauriello MC, Monfrecola A, Cameli N. Skin needling to enhance depigmenting serum penetration in the treatment of melasma. Plast Surg Int. 2011;2011:158241. doi: 10.1155/2011/158241. Epub 2011 Apr 7. PMID 22567235
- [Background] Goodman MP. Female genital cosmetic and plastic surgery: a review. J Sex Med. 2011 Jun;8(6):1813-25. doi: 10.1111/j.1743-6109.2011.02254.x. Epub 2011 Apr 14. PMID 21492397